CLINICAL TRIAL: NCT02814097
Title: A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effects of 4 Weeks Treatment With Subcutaneous Elamipretide on Left Ventricular Function in Subjects With Stable Heart Failure With Preserved Ejection Fraction
Brief Title: A Study to Evaluate the Effects of 4 Weeks Treatment With Subcutaneous Elamipretide on Left Ventricular Function in Subjects With Stable Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Collaborators: Charite University, Berlin, Germany (Other); SCIRENT Clinical Research and Science d.o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIHF-203; 2015-005615-32 (EudraCT Number)
Record Dates: First submitted 2016-06-08; First posted 2016-06-27 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; HFpEF; elamipretide; MTP-131; Bendavia™
MeSH Terms: conditions — Heart Failure | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 mg elamipretide (Experimental): 40 mg elamipretide once daily for 28 consecutive days
  Interventions: Drug: elamipretide
- Placebo (Placebo Comparator): Placebo once daily for 28 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: elamipretide — Subcutaneous injection of 40 mg elamipretide once daily for 28 consecutive days
  Other Names: MTP-131; Bendavia
  Arms: 40 mg elamipretide
Drug: Placebo — Subcutaneous injection of placebo administered once daily for 28 consecutive days
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study in subjects with stable heart failure with preserved ejection fraction (HFpEF) to evaluate the effects of 4 weeks treatment with subcutaneous MTP-131 (elampretide) on left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 and <80 years.
* Symptomatic heart failure (i.e. NYHA II or III) due to HFpEF for at least 6 months prior to study start
* Evidence of HFpEF: LVEF ≥45% and E/e´>10 and NT-pro-BNP >220 pg/ml (sinus rhythm) / > 600 pg/mL (atrial fibrillation)
* An exercise-induced increase in E/e' of at least 1.5 units during stress echocardiography assessment.
* Heart failure is considered to be stable, in the judgment of the investigator, and no hospitalization for HFpEF or changes in dose regimen of pharmacologic treatment for HF has occurred within 1 month prior to the Screening Visit.
* Treatment with appropriate pharmacologic therapy to manage underlying risk factors according to current guidelines.
* Women of childbearing potential must agree to use 1 of the following methods of birth control from the date they sign the ICF until two months after the last dose of study medication:

  a) Abstinence, b) surgically sterilized male partner, or c) barrier method And hormonal contraception
* Women of child-bearing potential must have a negative serum pregnancy test at baseline
* Willing and able to provide signed informed consent form (ICF) prior to participation in any study-related procedures

Exclusion Criteria:

* Probable alternative diagnoses that in the opinion of the investigator could account for the patient's symptoms e.g. severe pulmonary dysfunction or severe asthma
* LVEF <45% (at the moment of enrollment or in medical history)
* Coronary or peripheral revascularization procedures, valvular procedures, OR any major surgical procedure within 3 months prior to the Screening Visit.
* Acute coronary syndrome (ACS), stroke or transient ischemic attack (TIA) within 3 months prior to the Screening Visit.
* Uncontrolled hypertension defined as a systolic blood pressure (BP) >160 mm Hg or a diastolic BP >100 mm Hg on at least 2 consecutive readings that will require a change in anti-hypertensive treatment during the study period.
* Active cancer or undergoing chemotherapy within previous 6 months
* Total bilirubin >2x the upper limit of normal (ULN) in the absence of Gilbert's Syndrome (M. Meulengracht) and liver enzymes (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] and/or alkaline phosphatase) elevation >3xULN
* Estimated glomerular filtration rate <30 mL/min, by MDRD
* Known active drug or alcohol abuse within 1 year of the Screening Visit.
* Use of other investigational drugs at the time of enrolment, or within 30 days or 5 half-lives of enrolment
* Treatment with spironolactone or eplerenone for less than 3 months at study start
* Treatment with dabigatran
* Treatment with valsartan/sacubitril
* Female subjects who are pregnant, planning to become pregnant, or lactating.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Compare the delta in E/e' at rest exercise measured with echocardiography between the elamipretide and placebo groups | 4 weeks

SECONDARY OUTCOMES:
Compare the change at rest and during submaximal stress in LV systolic global longitudinal strain (GLS) between the elamipretide and placebo groups at the end of the 4-week treatment period | 4 weeks
Compare the change in 6-minute walking distance, between the elamipretide and placebo groups at the end of the 4-week treatment period | 4 weeks
Compare the change in NT-proBNP, between the elamipretide and placebo groups at the end of the 4-week treatment period | 4 weeks
Compare the percent of patients on elamipretide versus placebo presenting with TEAEs and SAEs, including changes in biomarkers of myocardial damage and changes in markers of renal function | 4 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (2):
  - Charite Universitatsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - German Heart Center, Berlin
- Serbia (7):
  - Clinical Centre of Serbia, Clinic for Cardiology, Belgrade
  - Clinical Hospital Center "Dr Dragiša Mišović-Dedinje", Department of Cardiology, Belgrade
  - Clinical Hospital Center "Zvezdara", Department of Cardiology, Belgrade
  - Clinical Hospital Center "Bežanijska Kosa", Department of Cardiology, Belgrade
  - Clinical Hospital Center "Zemun", Department of Cardiology, Belgrade
  - Institute for Cardiovascular Diseases Vojvodina, Clinic for Cardiology, Kamenitz
  - Clinical Center Niš, Clinic for Cardiology, Niš